CLINICAL TRIAL: NCT03734640
Title: Optimal Post Tpa-Iv Monitoring in Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Anderson (Other)
Collaborators: Genentech, Inc. (Industry); Johns Hopkins University (Other); The George Institute for Global Health, Australia (Other)
Responsible Party: Sponsor-Investigator, Craig Anderson, Executive Director, The George Institute for Global Health, China
Organization: The George Institute for Global Health, China (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPTIMISTmain
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke Patients Receiving Reperfusion Therapy

STUDY DESIGN:
Intervention Model Description: stepped wedge cluster randomized
Who Masked: Outcomes Assessor
Masking Description: Guardian consent for intervention as standard of care service provision. Outcome assessed by independent researcher blind to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guideline recommended standard monitoring (Placebo Comparator): vital signs (HR, BP) and neurological assessment (GCS and NIHSS) 15-30mins x 2 hours, 30mins x 6 hours, 1hourly x 16 hours in usual care monitoring environment
  Interventions: Other: Guideline recommended standard monitoring
- Low-intensity monitoring strategy (Active Comparator): vital signs (HR, BP) and neurological assessment (GCS and/or NIHSS) 15-30mins x 2 hours, 2hourly x 8 hours, 4hourly x 14 hours in a non-ICU ward
  Interventions: Other: Low-intensity monitoring strategy

INTERVENTIONS:
Other: Low-intensity monitoring strategy — Post-tpa patients will be monitored in a lower intensity with less vital status and neurological assessment
  Arms: Low-intensity monitoring strategy
Other: Guideline recommended standard monitoring — Post-tpa patients will be monitored in the usual care monitoring environment
  Arms: Guideline recommended standard monitoring

SUMMARY:
OPTIMISTmain is an investigator-initiated and conducted, international, multicentre, stepped wedge cluster randomized controlled trial comparing the effects of different intensities of nursing care monitoring for patients with acute ischemic stroke of mild severity and without critical care needs after IV-tPA.

DETAILED DESCRIPTION:
Research question: Patients receiving thrombolytic therapy (tissue plasminogen activator [tPA]) for acute ischaemic stroke (AIS), have been monitored with a high intensity schedule of vital signs and neurologic assessments, which often requires 1:1 nursing and/or admission in an intensive care unit (ICU) or similar ward for at least 24 hours after receiving tPA. Studies indicate that patients with mild degrees of AIS after tPA do not require such intensive monitoring, yet most stroke services continue to follow a practice recommended in guidelines based on the initial cautious evaluation of tPA in AIS over 20 years ago.

Design: Stepped-wedge cluster randomised design. With 3 groups and 4 phases. All groups starting with standard care and in each subsequent phase, groups I through III will switch to the intervention (low-intensity monitoring).

Study centers: This is a global study. Approximately 157 hospitals ('sites') in Australasia, Europe, South American, and North American regions, who are willing to accept the randomized intervention change and adhere to the protocol, collect a required minimum data set on patients over 7 days in hospital (or discharge or death, if sooner), and record any serious adverse event (SAE) during and at clinical outcome assessed at 90 days of follow-up of patients.

Consent/randomization: Hospitals will be eligible if they are using the proposed low-intensity nursing monitoring strategy. A stepped-wedge cluster randomized design has been chosen to avoid contamination, facilitate hospital-wide implementation, and maximize adherence, as the intervention under investigation is to become usual standard of care. The process of one direction (from control to intervention) is to facilitate the low intensity monitoring protocol being applied in clinical practice. The stepped-wedge design means that all hospitals will be randomly allocated to 3 groups: in phase 1, all hospitals will be observed under standard care 'control' conditions according to guideline recommended monitoring; in phase 2, the first cluster of hospitals (Group I) will start receiving the intervention (low-intensity), and then sequentially, Groups II and III will start receiving the interventional package in phase 3 and 4, respectively, so that by phase 4, all hospitals will have the intervention. Those hospitals in Group I are exposed to the intervention for longest time, and those in Group III, the shortest time.

In each phase, hospitals are to maintain a register of all thrombolyzed AIS patients, and to identify all those eligible for, or excluded from participating in the study. Hospitals are required to manage at minimum target of at least 10 consecutive thrombolyzed AIS patients who fulfill the eligibility criteria (presumed 50% of all thrombolyzed AIS patients) over each 4 month period. The recruitment number will vary from 10 to 30 patients, according to seasonal fluctuation and overall numbers of thrombolyzed AIS patients across hospitals. The target number and time limits for each phase will be pre-determined and agreed to with each hospital, to ensure an orderly completion of the study.

On average, for Group I, the time for initiation of the low-intensive intervention is 4 months after activation into phase 1 of the study; for Groups II and III, the time periods for initiation of the low-intensive intervention are 6 and 9 months, after activation, respectively. Data collection will occur at baseline, the first 24 hours, Day 7 (or death or time of hospital discharge, if earlier), and at 90 days (end of follow-up). Patients will be asked to consent to being contacted at some future date to examine long-term outcomes, according to available resources.

A senior executive officer at each center will act as a 'guardian', to provide consent at an institutional level for the intervention to be applied as a 'low risk' intervention to clusters of patients as part of routine care; and written informed consent is to be subsequently obtained from participants, or their approved surrogates, for collection of medical data and participation in the follow-up assessments Randomized allocation of intervention will be assigned by a statistician not otherwise involved in the study according to a statistical program stratified by the country of the site.

Sample size: The sample size required to detect a plausible treatment effect on a clinical outcome in a stepped-wedge trial (3 groups, 4 phases) is 157 hospitals, each recruiting an average of 80 patients (20 per phase), for a total of 12,394 AIS patients. The basis of this calculation is that the study is designed with 90% power (one-sided α = 0.025) to detect non-inferiority (non-inferiority OR margin is 1.25, presumed actual OR is 1.0; the proportion of a bad outcome [mRS 2-6] is 50%) of low-intensity monitoring on the primary outcome. Assuming a stepped-wedge trial of 3 groups and 4 phases, 157 hospitals are required to be randomized into 3 groups of 53 hospitals, each recruiting an average of 16 patients per phase, for a total of 9340 subjects. Assuming 10% with missing primary endpoint data and 5% with nonadherence to randomized treatment, the overall sample size increases to an average of 20 subjects per hospital per phase (i.e. total sample size of 12,394 AIS patients). Allowance will be made to include some very large hospitals (10%, 7) to recruit 50 patients per phase, and smaller hospitals (10%, 7) to recruit 8 patients per phase, in order to allow a broad range of hospitals with variable experience and systems of care for the management of AIS.

ELIGIBILITY:
Inclusion Criteria:

* adults (age ≥18 years);
* have received IV alteplase for AIS according to standard criteria;
* have a mild-moderate level of neurological impairment (e.g. score <10 on the NIHSS);
* stable and without any critical care needs at the end of the infusion of alteplase.

Exclusion Criteria:

* major neurological impairment;
* definite clinical contraindication or indication to either low-intensity or standard neurological monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4922 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
modified Rankin scale (mRS); shift analysis across full range of scores | day 90
  Physical function measured according to a 7 level categorical scale, where 0-1 indicates no or minimal symptoms, 2-5 indicates increasing levels of disability/dependencey, and 6=death

SECONDARY OUTCOMES:
frequency of major Symptomatic intracerebral hemorrhage | day 90
  intracerebral hemorrhage on brain imaging associated with significant neurological deterioration or death over 24 hours
Measures of hospital costs | day 90
  to allow economic analysis of treatment interventions at a country level
any serious adverse event during follow-up | Within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Craig S Anderson, MD PhD, Principal Investigator — The George Institute; Victor C Urrutia, MD, Principal Investigator — Johns Hopkins University
Locations (54):
- United States (20):
  - Centura St. Anthony Hospital, Lakewood, Colorado
  - Centura Littleton Adventist Hospital, Littleton, Colorado
  - University of Maryland Medical Center, Baltimore, Maryland
  - The John Hopkins Hospital, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Ascension Providence Hospital, Novi, Michigan
  - SSM Health DePaul Hospital, Bridgeton, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Renown Health, Reno, Nevada
  - University of Rochester Medical Center, Rochester, New York
  - Cone Health, Greensboro, North Carolina
  - OhioHealth Research Institute - Riverside Methodist Hospital, Columbus, Ohio
  - INTEGRIS Southwest Medical Center, Oklahoma City, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Penn State Health, Hershey, Pennsylvania
  - Inova Fairfax Hospital, Falls Church, Virginia
  - ThedaCare Regional Medical Center Appleton, Appleton, Wisconsin
- Australia (9):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Concord Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Public Hospital, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Chile (8):
  - Hospital de Puerto Montt, Port Montt, Los Lagos Region
  - Clinica Alemana de Santiago, Santiago, Santiago Metropolitan
  - Hospital del Pino, Santiago, Santiago Metropolitan
  - Hospital La Florida Dra. Eloisa Díaz, Santiago, Santiago Metropolitan
  - Hospital Padre Hurtado, Santiago, Santiago Metropolitan
  - Hospital Sótero del Rio, Santiago, Santiago Metropolitan
  - Hospital Base de Osorno, Osorno
  - Hospital Carlos Van Buren, Valparaíso
- Shenyang First People's Hospital, Shenyang, China
- Malaysia (3):
  - Hospital Universiti Sains Malaysia, Kota Bharu
  - Universiti Kebangssan Malaysia Medical Center, Kuala Lumpur
  - Hospital Pengajar Universiti Putra Malaysia (Hpupm), Serdang
- Mexico (2):
  - Instituto Nacional de Neurología y Neurocirugía Manuel Velasco Suarez, Mexico City
  - Hospital Regional ISSSTE de Puebla, Puebla City
- United Kingdom (11):
  - Addenbrookes Hospital, Cambridge
  - Countess of Chester Hospital, Chester
  - Royal Devon and Exeter Hospital, Exeter
  - Leicester Royal Infirmary, London
  - University College London Hospitals, London
  - Kings College Hospital, London
  - St George's University Hospitals, London
  - Luton and Dunstable University Hospital, Luton
  - Nottingham University Hospitals, Nottingham
  - Warnford Hospital, Oxford
  - Peterborough City Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
12 months after completion of the study, experienced researchers can seek a copy of the database through requests to the Research Office of The George Institute
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months after primary results publication
Access Criteria: Request with protocol to the Research Office of The George Institute

REFERENCES:
- [Derived] Xu L, Ouyang M, Atkins ER, Summers D, Sui Y, Johnson B, Billot L, Malavera A, Faigle R, Munoz-Venturelli P, Day D, Liu X, Li Q, Song L, Robinson TG, Gonzalez F, Urrutia-Goldsack F, Delcourt C, Nguyen HT, Ton MD, Liu H, Lindley RI, Arauz A, Mercado A, Wan Zaidi WA, Khatri P, Wang X, Urrutia VC, Jan S, Anderson CS. Low-Intensity Monitoring for Mild-to-Moderate Acute Ischemic Stroke Is Cost Saving: Economic Evaluation for OPTIMISTmain. Stroke. 2026 Jan 29. doi: 10.1161/STROKEAHA.125.053506. Online ahead of print. PMID 41608808
- [Derived] Anderson CS, Summers D, Ouyang M, Sui Y, Johnson B, Billot L, Malavera A, Faigle R, Munoz-Venturelli P, Day D, Liu X, Li Q, Song L, Robinson TG, Gonzalez F, Urrutia-Goldsack F, Iacobelli M, Montalbano M, Pruski A, Delcourt C, Durham AC, Ebraimo A, Van Ta HH, Ghosh P, Leonhardt-Caprio A, Nguyen HT, Ton MD, Jan S, Liu H, Lindley RI, Arauz A, Mercado A, Zaidi WAW, Khatri P, Wang X, Urrutia VC; OPTIMISTmain Investigators. Safety and efficacy of low-intensity versus standard monitoring following intravenous thrombolytic treatment in patients with acute ischaemic stroke (OPTIMISTmain): an international, pragmatic, stepped-wedge, cluster-randomised, controlled non-inferiority trial. Lancet. 2025 May 31;405(10493):1909-1922. doi: 10.1016/S0140-6736(25)00549-5. Epub 2025 May 21. PMID 40412428